CLINICAL TRIAL: NCT00295997
Title: Non-myeloablative Allogeneic Stem Cell Transplantation With Match Unrelated Donors for Treatment of Hematologic Malignancies and Renal Cell Carcinoma and Aplastic Anemia
Brief Title: Donor Stem Cell Transplant in Treating Patients With Hematologic Cancer, Metastatic Kidney Cancer, or Aplastic Anemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000463522; UCSF-01251; UCSF-H5010-19585-05; UCSF-2101
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2007-04

CONDITIONS: Chronic Myeloproliferative Disorders; Kidney Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; essential thrombocythemia; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; polycythemia vera; previously treated myelodysplastic syndromes; recurrent adult acute myeloid leukemia; prolymphocytic leukemia; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; refractory chronic lymphocytic leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; stage II multiple myeloma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III multiple myeloma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent renal cell cancer; stage IV renal cell cancer; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent adult acute lymphoblastic leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Kidney Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Thrombocythemia, Essential; Leukemia, Myelomonocytic, Juvenile; Polycythemia Vera; Leukemia, Myeloid, Acute; Leukemia, Prolymphocytic; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Carcinoma, Renal Cell | interventions — Antilymphocyte Serum; Filgrastim; Busulfan; Cyclophosphamide; fludarabine phosphate; Methotrexate; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Biological: graft-versus-tumor induction therapy
Biological: therapeutic allogeneic lymphocytes
Drug: busulfan
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: methotrexate
Drug: mycophenolate mofetil
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy before a donor stem cell transplant using stem cells that closely match the patient's stem cells, helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving antithymocyte globulin before transplant and cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well a donor stem cell transplant works in treating patients with hematologic cancer, metastatic kidney cancer, or aplastic anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the treatment-related mortality (TRM) rate at 100 days in patients with hematologic malignancy, metastatic renal cell carcinoma, or aplastic anemia undergoing nonmyeloablative allogeneic stem cell transplantation using matched unrelated donors.

Secondary

* Determine the TRM at 12 months in patients treated with this regimen.
* Determine the 6-month engraftment rate in patients treated with this regimen.
* Determine 1-year overall survival of patients treated with this regimen.

OUTLINE:

* Nonmyeloablative preparative regimen: Patients receive fludarabine IV over 30 minutes on days -7 to -3, busulfan* IV over 6 hours on days -4 and -3, and anti-thymocyte globulin IV over 6-10 hours on days -4 to -1.

NOTE: *Patients with aplastic anemia receive cyclophosphamide IV over 2 hours on days -6 to -3 instead of busulfan.

* Allogeneic stem cell reinfusion: Patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation on day 0. Patients then receive filgrastim (G-CSF) subcutaneously daily beginning on day 7 and continuing until blood counts recover.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive tacrolimus orally twice daily or IV continuously beginning on day -2 and continuing for approximately for 6-12 months after transplantation. Patients also receive mycophenolate mofetil orally or IV twice daily on days 0 to 60 and methotrexate IV on days 1, 3, 6, and 11**.

NOTE: **Patients with aplastic anemia receive methotrexate IV on days 1, 3, and 6 (not day 11).

* Donor lymphocyte infusion (DLI): After day 180, patients with no evidence of active GVHD may receive DLI. A second DLI may be infused > 8 weeks after the first in the absence of disease response or GVHD.

After completion of study treatment, patients are followed periodically for at least 2 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Aplastic anemia not responsive to immunosuppressive therapy
  * Metastatic renal cell carcinoma
  * Hematologic malignancy, including any of the following:

    * Acute myeloid leukemia (AML)* not curable with chemotherapy and meeting any of the following criteria:

      * AML with high-risk cytogenetic abnormalities (e.g., -7, -7q, -5, -5q, complex, Philadelphia chromosome-positive [Ph+])
      * AML evolved from prior myelodysplasia
      * AML secondary to prior chemotherapy
      * Failed to achieve remission
      * In second or subsequent remission NOTE: *Marrow blasts < 10%- can be achieved by chemotherapy
    * Myelodysplasia* with any of the following high-risk features:

      * Adverse cytogenetics (-7, 7q, -5, -5q, complex)
      * Excess blasts
      * Prior conversion to AML
      * Severe cytopenias with absolute neutrophil count < 500/mm^3 or platelet count < 20,000/mm^3 NOTE: *Marrow blasts < 10%- can be achieved by chemotherapy
    * Acute lymphoblastic leukemia (ALL)* not curable with chemotherapy and meeting any of the following criteria:

      * High-risk cytogenetics (Ph+, 11q23 abnormalities, monosomy 7)
      * More than 1 induction course required to achieve remission
      * Failed to enter remission
      * In second or subsequent remission NOTE: *Marrow blasts < 10 %
    * Chronic lymphocytic leukemia (CLL) with high-risk features, including any of the following:

      * Refractory to initial or subsequent therapy
      * Progression after initial response to therapy
      * Prolymphocytic morphology
    * Follicular lymphoma with any of the following high-risk features:

      * Refractory to initial or subsequent therapy
      * Progression after response to initial therapy
      * Has ≥ 3 International Prognostic Index (IPI) risk factors
    * Multiple myeloma

      * Stage II-III disease confirmed at diagnosis or after initial progression
    * Other lymphoma that has failed to respond to primary therapy, progressed, or recurred after prior therapy, including any of the following:

      * Diffuse large cell lymphoma
      * Mantle cell lymphoma
      * Hodgkin's lymphoma
    * Myeloproliferative disease with evidence of disease acceleration, including any of the following:

      * Myelofibrosis
      * Polycythemia vera
      * Essential thrombocythemia
    * Chronic myeloid leukemia (CML) that failed to be controlled by imatinib mesylate
* Disease must be stable or responding to therapy
* No rapid progression of malignant disease

  * Expected time to disease progression > 12 weeks
* Not eligible for autologous stem cell transplantation
* Matched unrelated donor available

  * 9/10 HLA matched, including HLA-A, -B, -C, -DR, and -DQ

PATIENT CHARACTERISTICS:

* Creatinine < 2.0 mg/dL
* Creatinine clearance > 40 mL/min
* Bilirubin < 3 mg/dL

  * Elevated total bilirubin due to Gilbert's disease allowed if direct bilirubin is normal
* AST < 4 times upper limit of normal
* Hepatitis C or B allowed provided bilirubin and AST are normal
* Cardiac ejection fraction > 30%
* DLCO > 40% of predicted
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled active infection requiring ongoing antibiotic treatment
* No poor performance status
* No poor organ function

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior stem cell or bone marrow transplantation allowed

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Charles A. Linker, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina